CLINICAL TRIAL: NCT02413411
Title: Race and Preference for Knee Replacement: A Patient-Centered Intervention
Acronym: REPAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1-RO1-AR-054474-5; 1R01AR054474 (NIH)
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Knee Osteoarthritis
Keywords: Arthroplasty; Osteoarthritis; Replacement; Intervention
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DA/MI Intervention (Experimental): Patients randomized to the DA/MI intervention arm will be shown a decision aid video entitled, Treatment Choices for Knee Osteoarthritis. Following the viewing of the decision aid video, the participant will be engaged in a motivational interview by the research study interventionist.
  Interventions: Behavioral: DA/MI Intervention
- Attention Control (Active Comparator): Patients randomized to the attention control arm will receive an educational program (an NIH-developed booklet) that summarizes how to live with knee OA but does not specifically mention joint replacement. This booklet provides examples of exercises one could do to improve pain and reduce stiffness from knee OA.
  Interventions: Behavioral: an educational program (an NIH-developed booklet)

INTERVENTIONS:
Behavioral: DA/MI Intervention — Patients randomized to the DA/MI intervention arm will be shown a decision aid video entitled, Treatment Choices for Knee Osteoarthritis. Following the viewing of the decision aid video, the participant will be engaged in a motivational interview by the research study interventionist.
  Arms: DA/MI Intervention
Behavioral: an educational program (an NIH-developed booklet)
  Arms: Attention Control

SUMMARY:
A randomized, controlled design will be utilized to examine and compare the effectiveness of the proposed educational intervention, which includes a combination of an educational decision aid and motivational interviewing with attention control on select key patient-centered and process of care outcomes. The study sample will consist of approximately 450 African-American patients with osteoarthritis of the knee. Patients will be recruited from the University of Pennsylvania Health System and the Philadelphia VA Medical Center and will be randomized to one of the two study arms.

The immediate goal of this randomized controlled trial is to assess the effect of a high-quality, evidence-based, patient-centered educational intervention supplemented with targeted counseling (motivational interviewing) on African American patient preferences, expectations, and the likelihood of achieving a referral for surgical evaluation. The long-term goal of this research is to widely implement a patient-centered educational intervention targeting African Americans who are potential candidates for joint replacement, in a national effort to reduce and ultimately eliminate racial disparities in the utilization of this effective treatment option.

Study Aim:To examine the effect of the knee osteoarthritis Decision Aid (DA)/Motivational Interviewing (MI) intervention on orthopedic surgery referral rates for African American (AA) patients. Hypothesis: Compared to attention control, the DA/MI intervention will lead to higher orthopedic surgery referral rates for AA patients.

Secondary aim: To examine the effect of the DA/MI intervention on the rate of knee replacement receipt among AA patients. Hypothesis: AA patients randomized to receive the intervention will have higher rates of knee replacement compared to those in the attention control group.

DETAILED DESCRIPTION:
The study involves a baseline questionnaire, educational intervention, primary care follow-up phone call questionnaire (approximately 2 weeks after primary care appointment), and follow-up questionnaires by phone calls at 3 months and 1 year. All eligible, consented patients will complete the baseline questionnaire, conducted by a REPAIR research staff member. The baseline questionnaire will include the following instruments that have been field-tested by our team in previous and ongoing studies: 1.) Willingness to Consider Joint Replacement Question 2.) Knowledge Regarding Knee OA and Joint Replacement (developed by The Foundation for Informed Medical Decision Making) 3.) Hospital for Special Surgery Knee Expectations Survey 4.) Socioeconomic Survey 5.) Access to Health Care, Charleson Comorbidity Index 6.) Quality of Life SF-12v2. This survey can be done over the phone or in person. It should take approximately 30-40 minutes. At the completion of the baseline questionnaire, patients will be randomized into either study Decision Aid (DA) supplemented by motivational interview (MI) (hereafter referred to as DA/MI intervention) arm or the attention control arm. Patient appointments for the DA/MI intervention or attention control activity will be scheduled to occur 2 weeks prior to the patients next primary care appointment (up to the date of the appointment). The DA/MI intervention (referred to as an information session in patient material) will be completed by a REPAIR research study interventionist (the interventionist will not administer the baseline assessment). In the intervention arm, patients will be shown a decision aid video entitled, Treatment Choices for Knee Osteoarthritis. Following the viewing of the decision aid video, the participant will be engaged in a motivational interview by the research study interventionist.The completion time for the educational intervention will vary from 30 to 80 minutes. The attention control arm will be conducted by the REPAIR research staff. Patients will be given written educational material adapted from the NIH/NIAMS publication Osteoarthritis to review at his/her leisure.The completion time for the attention control arm is approximately 10 minutes. Follow-up procedures will occur at the following time points: 1.) approximately 2 weeks after the participants primary care appointment, 2.) 3-months post intervention, 3.) 12-months post intervention, and 4.) medical chart assessment. All followup procedures will be administered by a REPAIR research team member that was not involved in the educational intervention. Participants in both the DA/MI intervention and the attention control will complete a primary care follow-up survey approximately 2 weeks following the patients next primary care appointment. This survey will be comprised of the following: 1.) Willingness to consider joint replacement question 2.) Hospital for Special Surgery Knee Expectations Survey 3.) Knowledge Regarding Knee OA and Joint Replacement 4.) Communication questions regarding who the patient talked to about their knee pain and/or the intervention. The follow-up will take 10-15 minutes to complete, and will be administered preferably by phone. Participants in both the DA/MI intervention and the attention control will complete a 3-month follow-up (completed approximately 3 months post intervention) survey over the phone. This survey will be comprised the same as the primary care followup survey. This survey will take 10-15 minutes to complete. Lastly, participants in both the DA/MI intervention and the attention control will complete a 12-month follow-up (completed approximately 12 months post intervention) survey over the phone. The survey will be comprised of the following: Willingness to consider joint replacement, Hospital for Special Surgery Knee Expectations Survey, Knowledge Regarding Knee OA and Joint Replacement, and a survey regarding referrals to orthopedics and for joint replacement. At the time of the 12-month follow-up, the patients medical record will be accessed to check for a referral to orthopedics and a joint replacement procedure.

ELIGIBILITY:
Inclusion Criteria:

* African American primary care patients
* Age 50 or older
* Chronic, frequent knee pain based on the NHANES questions
* Moderate to sever knee osteoarthritis based on WOMAC index score greater than or equal to 39 or positive answer to knee treatment questions
* Radiographic evidence of knee osteoarthritis

Exclusion Criteria:

* Prior history of any major joint replacement
* Terminal illness (e.g. end stage cancer)
* Physician-diagnosed inflammatory arthritis (i.e., rheumatoid arthritis, connective tissue disease, ankylosing spondylitis, or other seronegative sypondylarthoplasty.)
* Contra-indications to replacement surgery (e.g., lower extremity paralysis as a result of stroke.)
* Prosthetic leg
* Cognitive impairment (e.g., dementia)
* No home telephone service

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Referral to knee joint replacement | 12-months post-intervention
  Referral to knee joint replacement will be assessed for all patients 12 months post-intervention initially through telephone survey and then validated by medical record review

SECONDARY OUTCOMES:
Receipt of knee joint replacement | 12-months post-intervention
  Receipt of knee joint replacement will be assessed for all patients 12-months post-intervention initially through telephone survey and then validated by medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Said A Ibrahim, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States